CLINICAL TRIAL: NCT03570281
Title: Edoxaban for the Treatment of Coagulopathy in Patients With Active Cancer and Acute Ischemic Stroke: a Pilot Study. (ENCHASE Study)
Acronym: ENCHASE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Oh Young Bang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2017-11-163-007
Record Dates: First submitted 2018-05-14; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Correction of Cancer-related Coagulopathy With Novel Oral Anticoagulant (Edoxaban)
Keywords: cancer-related stroke; coagulopathy; D-dimer; Edoxaban; enoxaparine
MeSH Terms: conditions — Hemostatic Disorders | interventions — edoxaban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edoxaban group (Experimental): Edoxaban, per oral, 60mg qd (may consider reduced dose to 30mg qd in patients with proper clinical reason by attending physician, estimated creatinine clearance of 30 to 50 ml per minute, a body weight of 60 kg or less, or the concomitant use of verapamil or quinidine), for 90 days.
  Interventions: Drug: Edoxaban
- Enoxaparin group (Active Comparator): Enoxaparin, subcutaneous injection, 1mg/kg BID (may consider reduced dose to 1mg/kg qd in patients with proper clinical reason by attending physician, Creatinine clearance <30 mL/min), for 90 days.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Edoxaban — Edoxaban, per oral, 60mg qd (may consider reduced dose to 30mg qd in patients with proper clinical reason by attending physician, estimated creatinine clearance of 30 to 50 ml per minute, a body weight of 60 kg or less, or the concomitant use of verapamil or quinidine), for 90 days.
  Arms: Edoxaban group
Drug: Enoxaparin — Enoxaparin, subcutaneous injection, 1mg/kg BID (may consider reduced dose to 1mg/kg qd in patients with proper clinical reason by attending physician, Creatinine clearance <30 mL/min), for 90 days.
  Arms: Enoxaparin group

SUMMARY:
Purpose: Cancer-related hypercoagulability plays an important role in the development of cancer-related stroke. With rapidly aging population and increasing cancer prevalence, cancer related stroke has become an important stroke subtype. Recent studies suggest that hypercoagulability is associated with poor prognosis and effective correction of coagulopathy maybe protective for survival in cancer related stroke patients. Optimal strategies to correct coagulopathy in cancer stroke patient remains to be determined. Currently, the use of low molecular-weighted heparin is recommended in these patients, but non-vitamin K oral anticoagulants (NOACs) could be safe alternative without the need for injection subcutaneously. Furthermore, NOACs could be an optimal treatment strategy for cancer-related stroke in terms of correcting coagulopathy with less injection related complication (ex. pain and infection) compared to Enoxaparin.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years old
* Acute cerebral infarction within 30 days of symptom onset was confirmed by diffusion-weighted brain magnetic resonance imaging (DWI)
* Cancer-related stroke, not diagnosed with other classic (arteriosclerosis, cardioembolicm, small-vessel occlusion, etc.) cerebral infarction, within six months of diagnosis, chemotherapy, surgery for cancer.
* with informed consent from the patient or next-of-kin, When the subject becomes able to decide whether to participate in the study, the researcher acquires further consent directly from the subject.

Exclusion Criteria:

* Patients with primary intracranial malignancy
* Patients with classic causes of cerebral infarction
* Patients with infectious or immunological disease that may affect blood D-dimer levels
* Patients whose cerebral infarction is thought to be caused by tumor (vascular occlusion due to tumor tissue)
* Patients who can not use anticoagulants with thrombocytopenia (platelet <50,000), anemia (hemoglobin <8)
* Decreased renal function (creatine clearance <15 mL / mim)
* Patients who received intravenous tissue plasminogen activator
* Patients with uncontrolled severe hypertension
* Patients who received prosthetic heart valve replacement requiring anticoagulation
* Patients with moderate to severe mitral stenosis
* Pulmonary embolism requiring hemodynamically unstable or thrombolysis or pulmonary embolization
* Pregnant and lactating women
* Patients who are hypersensitive to the major component or constituent of the test drug
* Patients with liver diseases associated with blood clotting disorders and clinically significant bleeding risks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
D-dimer change | 7 days after treatment
  interval change of serum D-dimer level between day 0 and 7

SECONDARY OUTCOMES:
Surrogate endpoint | 7 days after treatment
  number of micro-embolic signal detected by transcranial doppler
Functional outcome | 90 days after enrollment
  modified Rankin scale at 90 days, from 0 to 6, higher is worse
Incidence of Treatment-Emergent Adverse Events [symptomatic intracerebral hemorrhage] | 90 days after enrollment
  symptomatic intracerebral hemorrhage major bleeding all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chung JW, Hwang J, Kim HJ, Seo WK, Ahn MJ, Saver JL, Bang OY. Edoxaban for the treatment of hypercoagulability and cerebral thromboembolism associated with cancer: A randomized clinical trial of biomarker targets. Int J Stroke. 2024 Jul;19(6):645-653. doi: 10.1177/17474930241239266. Epub 2024 Mar 21. PMID 38429253